CLINICAL TRIAL: NCT06227351
Title: Accuracy of Completely Versus Partially Limiting Computer Guided Zygomatic Implant Placement. a Randomized Controlled Study
Brief Title: Completely Versus Partially Guided Zygomatic Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mohamed Kamal Hassan Ghallab, Teaching assistant in the Department of Oral and Maxillofacial Surgery, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Zygomatic Implant
Record Dates: First submitted 2024-01-16; First posted 2024-01-26 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-04

CONDITIONS: Maxillary Deficiency; Alveolar Bone Loss
Keywords: zygomatic implant; guided surgery; deficient maxilla
MeSH Terms: conditions — Retrognathia; Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized (1:1) clinical trial study formed of 2 competitive groups where 12 implants will be placed in 2 groups (6 for each group) to compare the accuracy of completely limiting computer generated surgical three-dimensional guide versus partially limiting computer generated surgical three-dimensional guide during placement of zygomatic implants in patients with atrophic maxillae.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- completely limiting computer generated surgical three-dimensional guide (Active Comparator): patients in this group will receive zygomatic implant placed in a completely fully guided technique using surgical guide,keys and sleeves.
  Interventions: Procedure: completely limiting computer generated surgical three-dimensional guide
- Partially limiting computer generated surgical three-dimensional guide (Active Comparator): patients in this group will receive zygomatic implant placed in a partially guided technique using surgical guide.The first drill only will be used with the guide then the guide will be removed and the whole procedure with the remaining drills will be completed in a free hand technique.
  Interventions: Procedure: Partially limiting computer generated surgical three-dimensional guide

INTERVENTIONS:
Procedure: completely limiting computer generated surgical three-dimensional guide — Long mid-crestal incision from the right to the left maxillary tuberosity and raising a full thickness flap to expose the maxilla up to the fronto-zygomatic notch.
  According to the zygoma anatomy-guided approach classification and previously planned surgery using Cone beam C.T lateral window and sinus foor lifting will be decided to be done or not.
  After securing the surgical templates in its proper position, sequential osteotomy drilling will be performed in a steady in and out movement under copious sterile saline irrigation.The drills will be entering the maxilla palatally and puncturing the alveolar crest to reach the buccal side.The drills will be visualized through the bony window created until it reaches the zygomatic bone.Sequential drills with the uses of guided tubes,sleeves and keys will be used to guarantee that the implant have been placed in a fully completely guided manner.Afterwards the zygomatic implants will be placed.
  Arms: completely limiting computer generated surgical three-dimensional guide
Procedure: Partially limiting computer generated surgical three-dimensional guide — Long mid-crestal incision from the right to the left maxillary tuberosity and raising a full -thickness flap to expose the maxilla up to the fronto-zygomatic notch.
  According to zygoma anatomy-guided approach classification and previously planned surgery using cone beam C.T.lateral window and sinus floor lifting will be decided to be done or not.After securing the surgical templates,The first drill only will be used using the guide then it will be removed and the other drills will be completed in a free hand without the use of guide to guarantee that the implant will be placed in partially guided manner.Afterwards the zygomatic implants will be placed.
  Arms: Partially limiting computer generated surgical three-dimensional guide

SUMMARY:
The aim of study is evaluation of accuracy of completely versus partially limiting computer generated surgical three-dimensional guides during placement of zygoma implants in patients with atrophic maxillae.

DETAILED DESCRIPTION:
According to World Oral Health Organization (WHO), losing teeth and arch edentulism is the result of a life long history of oral diseases like advanced dental caries and severe periodontal disease. Complete tooth loss estimated global average prevalence is 7% among people aged 20 years and 23% among people aged 60 years or older. Tooth loss lead to bone resorption in all direction.

Non-grafting solutions have been developed to reduce risks, morbidity, and treatment time. These types of treatment are often preferred by patients, considering that they may minimize total treatment time and have less morbidity than staged procedures of grafting solutions.One of non-grafting solutions is the zygomatic implants.

Zygomatic implants have shown improved clinical results compared with bone grafting in compromised maxillary bone.But the same as any surgical procedure, placing zygomatic implants has potential complication, such as: oro-antral communication, paresthesia or altered sensation of the infra orbital nerve also penetration of the orbital cavity may occur. In order to achieve the optimal position of zygomatic implant, computer-based planning has been introduced with the use of surgical guides.

Surgical guides are classified according to design concepts for fabrication of surgical guide to non-limiting, partially limiting design and complete limiting. In partially limiting design,the first drill is used then the surgical guide is removed and the osteotomy and implant placement are completed in freehand while in complete limiting design all the instruments used in surgical procedure during implant placement are restricted.

In literature, there is low evidence of using partially guided surgery for zygomatic implant and also of comparing the two designs with each other. the aim of study is evaluation of accuracy of completely versus partially limiting computer generated surgical three-dimensional guides during placement of zygoma implants in patients with atrophic maxillae.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years.
2. Patients with severe alveolar bone atrophy in posterior maxilla (residual alveolar crest less than 4 mm in height, in the area immediately distal to the canine pillar).

Exclusion Criteria:

1. Patients with systemic conditions contra-indicating general anesthesia.
2. Patients with conditions contraindicating implant placement (e.g.: radiation to the head and neck, intra-venous bisphosphonates, uncontrolled Diabetes mellitus).
3. Patients with acute maxillary sinus infection or maxillary sinus cyst.
4. Restricted mouth opening (less than 3 cm inter-arch distance anteriorly).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Implant position | one week after the surgery.
  Comparing the position of implant post-operatively with the virtual planning pre-operatively.

SECONDARY OUTCOMES:
Surgery duration | from the start of surgery to the completion of surgery.
  By calculating the time from the start of surgery till the end of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum university, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No